CLINICAL TRIAL: NCT02921607
Title: Development of Scalable New Model(s) Focused on Care Co-ordination and Care Provision for Medically Complex, Co-morbid Chronic Disease Patient Segments Focusing on Heart Failure
Status: Completed | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Collaborators: ResMed (Industry); Boston Scientific Corporation (Industry); Cardiomark (Unknown)
Responsible Party: Sponsor
Other Study IDs: PHT/2016/16
Record Dates: First submitted 2016-09-21; First posted 2016-10-03 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational: One group - all participants will be completing questionnaires and will be followed up with three months post discharge.
  Interventions: Other: Observational group

INTERVENTIONS:
Other: Observational group — Participants will be asked to complete a questionnaire prior to discharge and 3 months later to follow up

SUMMARY:
The goal is to define a set of clinical pathways for heart failure patients, reflecting the period from prior to admission to the post-discharge period following hospitalisation, under the current system that exists at the two clinical sites [as mentioned previously, the main site is at St Vincent's University Hospital in Dublin, but to ensure generalizability the project team will also carry out similar work Portsmouth Hospital, United Kingdom]. These pathways have been drawn up using the experience of the clinical investigators, using an interactive workshop approach and a pilot study.

1. Pre-Admission Pathway
2. Emergency Department Pathway
3. In-Hospital management Pathway
4. Pre-discharge Pathway
5. Post-Discharge Pathway

During identification of these pathways, the research team identified the settings/personnel that require study to more fully comprehend the methods, strengths and weaknesses of the present processes. Study activities are focused on two aspects of the patient journey, immediately before discharge and three months post discharge during the outpatient phase.

DETAILED DESCRIPTION:
Heart failure is a significant public health issue with a prevalence of over 2%, and is among the leading causes of hospital admission worldwide, particularly in those over-65 years. Patients with heart failure frequently require acute hospitalisation and are at increased risk of mortality (more than half of heart failure patients will die within five years of initial diagnosis, American Heart Association). The high hospital admission rate and readmission reduce quality of life and significantly drive up the costs of health care provision for these patients. Moreover, there is a high variability in the reported readmission rates across institutions and countries, indicating that the structure of health care delivery is variable and of significant importance to outcome in this population. This study sets out to investigate the most clinically effective and cost- efficient method of delivering care to patients with heart failure focusing on the phase immediately before hospital admission, the hospital stay and the immediate discharge period, through analysis of the current standards of practice in both Ireland and the United Kingdom.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and above.
* With or without an established community diagnosis of heart failure.
* Admitted to the hospital through the Emergency Department or directly to the cardiology wards, for management of a primary problem/complaint of Acute Decompensated Heart Failure.
* Able and willing to provide written, informed consent.

Exclusion Criteria:

* Patients who present with primary non-heart failure presentation who may/may not have a secondary problem with heart failure, or stable heart failure not contributing to the present illness will be excluded.
* Also excluded will be those who cannot provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute decompensated heart failure
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-09; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Change in patient/carer questionnaire | Baseline data and three month post discharge
  to determine the extent to which the patient's day to day life is affected by heart failure. Also to determine the carer's level of involvement as a care giver and their opinion of the treatment/pathway

CONTACTS AND LOCATIONS:
Overall Officials: Paul Kalra, Study Director — Portsmouth Hospitals NHS Trust; Ken McDonald, Study Chair — St Vincent's University Hospital, Ireland
Locations (1):
- Portsmouth Hospitals NHS Trust, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Participant data will be shared in an anonymized form as part of a larger database and in a collaborative fashion.